CLINICAL TRIAL: NCT02920905
Title: Atracurium Mixed With Magnesium Sulfate Versus Atracurium Alone as Adjuvant to Lidocaine in Intravenous Regional Anesthesia
Brief Title: Atracurium Mixed With Magnesium Sulfate Versus Atracurium Alone as Adjuvant to Lidocaine in IVRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shimaa mamdouh mekkawy, resident doctor at anesthesia and ICU ,Assiut Univesity, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Li,atr,mg in ivra
Record Dates: First submitted 2016-08-25; First posted 2016-09-30 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Atracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- lidocaine (Experimental): • Patients in group A will receive 3 mg/kg of lidocaine 2% diluted with saline to a total volume of 40 ml.
  Interventions: Drug: Lidocaine
- lidocaine & atracurium (Experimental): • Patients in group B receive 3 mg/kg of lidocaine 2% + 2 mg atracurium diluted with saline to a total volume of 40 ml.
  Interventions: Drug: Lidocaine; Drug: atracurium
- lidocaine & atracurium & Mg sulphate (Experimental): • Patients in group C will receive 3 mg/kg of lidocaine 2% + 2 mg atracurium mixed with 10 mg /kg magnesium sulphate diluted with saline to a total volume of 40 ml.
  Interventions: Drug: Lidocaine; Drug: atracurium; Drug: Mg sulphate

INTERVENTIONS:
Drug: Lidocaine — Two intravenous cannulae will be placed; one in a vein on the dorsum of the hand to be operated (22 gauge) and the other in the opposite hand. A double tourniquet will be positioned on the upper arm of the hand to be operated. Arm will be elevated for 2 min.
  Circulatory isolation of arm will be confirmed by inspection of the color of the limb, absence of radial pulse and loss of pulse oximetry tracing in the ipsilateral index finger. The upper (proximal) tourniquet will then be inflated to a pressure of 100 mmHg above the systolic blood pressure of the patient. The anesthetic solution will be prepared by an observer and will be given over a period of 90 seconds.
Drug: atracurium — Two intravenous cannulae will be placed; one in a vein on the dorsum of the hand to be operated (22 gauge) and the other in the opposite hand. A double tourniquet will be positioned on the upper arm of the hand to be operated. Arm will be elevated for 2 min.
  Circulatory isolation of arm will be confirmed by inspection of the color of the limb, absence of radial pulse and loss of pulse oximetry tracing in the ipsilateral index finger. The upper (proximal) tourniquet will then be inflated to a pressure of 100 mmHg above the systolic blood pressure of the patient. The anesthetic solution will be prepared by an observer and will be given over a period of 90 seconds.
  Arms: lidocaine & atracurium; lidocaine & atracurium & Mg sulphate
Drug: Mg sulphate — Two intravenous cannulae will be placed; one in a vein on the dorsum of the hand to be operated (22 gauge) and the other in the opposite hand. A double tourniquet will be positioned on the upper arm of the hand to be operated. Arm will be elevated for 2 min.
  Circulatory isolation of arm will be confirmed by inspection of the color of the limb, absence of radial pulse . The upper (proximal) tourniquet will then be inflated to a pressure of 100 mmHg above the systolic blood pressure of the patient. The anesthetic solution will be prepared by an observer and will be given over a period of 90 seconds.
  Arms: lidocaine & atracurium & Mg sulphate

SUMMARY:
The present clinical study will be undertaken to compare study between the effect of atracurium with lidocaine versus addition of magnesium sulphate to the same doses with lidocaine administrated alone in IntraVenous Regional Anaesthesia to access motor block, sensory block, tourniquet pain and post operative analgesia .Also assessment of patient and surgeon satisfaction .

DETAILED DESCRIPTION:
patients will be divided randomly into three groups (A, B, C) of 25 each, according to computer generated table of random numbers.

* Patients in group A will receive 3 mg/kg of lidocaine 2% diluted with saline to a total volume of 40 ml.
* Patients in group B receive 3 mg/kg of lidocaine 2% + 2 mg atracurium diluted with saline to a total volume of 40 ml.
* Patients in group C will receive 3 mg/kg of lidocaine 2% + 2 mg atracurium mixed with 10 mg /kg magnesium sulphate diluted with saline to a total volume of 40 ml.

Onset of sensory block will be assessed by a pin prick performed at 1 minute interval in the dermatomal sensory distribution of the medial and lateral ante brachial cutaneous, ulnar, median and radial nerves. Sensory block onset time will be recorded as time elapsed from injection of drug to sensory block achieved in all dermatomes.Onset of motor block will be assessed by asking the subject to flex and extend his/her wrist and fingers. Monitoring of motor block will be assessed by Modified Bromage Score . Complete motor block will be recorded when no voluntary movement will be possible.

At the end of surgery, the tourniquet will be deflated by a cyclic deflation technique and recording this :

* Sensory block recovery time
* Motor block recovery time
* Mean arterial pressure (MAP),
* heart rate (HR)
* visual analogue scale (VAS) will be recorded at 0, 15 min , 1, 6, 12, and 24 h.
* The time to first analgesic requirement will be recorded (the time elapsed from tourniquet release until first patient request for analgesic).

Patient and surgeon satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Short procedures (less than 2 hours).
* Cooperative patients.

Exclusion Criteria:

* Patients with sickle cell anemia.
* History of drug allergy.
* Raynaud's disease.
* Scleroderma.
* Myasthenia gravis.
* Cardiac disease.
* Diabetes mellitus.
* Peptic ulcer.
* Gastritis.
* Liver or renal insufficiency.
* Patients with history of convulsions .

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia | 24 hour
  postoperative analgesia measured by VAS of 0-10 (0= no pain and 10=Worst pain imaginable ) during the first 24 hours

SECONDARY OUTCOMES:
The onset and recovary times of sensory and motor block , first analgesic request , tourniquet pain ,side effects of study drugs , and quality of anesthesia assessed by patients and surgeons | 24 hours
  Onset of sensory block assessed by pinbrick of the arm . Onset of motor block will be assessed by asking the subject to flex and extend his/her wrist and fingers. Monitoring of motor block will be assessed by Modified Bromage Score . Complete motor block will be recorded when no voluntary movement will be possible.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Abbas Youssef, Prof, Study Director — Assiut University; . Ola Mahmoud Wahba, Ass Prof, Study Director — Assiut University; Ghada Mohammad Abo Elfadl, Lecturer, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assiut University Hospital, Asyut
  - Asyut

IPD SHARING:
Plan to Share IPD: Undecided